CLINICAL TRIAL: NCT01073696
Title: A Phase I Study to Evaluate the Effect of External Heat on the Pharmacokinetics of a Transdermal Granisetron Patch in Healthy Subjects
Brief Title: Effect of External Heat on a Transdermal Granisetron Patch in Pharmacokinetics (PK) of Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Kyowa Kirin Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 392MD/43/C; 2009-017036-40 (EudraCT Number)
Record Dates: First submitted 2010-02-16; First posted 2010-02-23 (Estimated); Last update posted 2024-06-17 (Actual); Status verified 2024-06

CONDITIONS: Healthy
Keywords: Sancuso; granisetron; Pharmacokinetics

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- granisetron IV (Active Comparator)
  Interventions: Drug: granisetron IV
- granisetron patch (Experimental)
  Interventions: Drug: granisetron patch

INTERVENTIONS:
Drug: granisetron IV — IV
  Arms: granisetron IV
Drug: granisetron patch — patch
  Arms: granisetron patch

SUMMARY:
The purpose of this study is to determine the effect of heat applied to a granisetron transdermal patch in healthy subjects.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male or female subjects aged ≥ 18 and ≤ 45 years at screening. Subjects must demonstrate understanding of the purposes and risks of the study and agree to follow the restrictions and schedule of study procedures, as evidenced by voluntary written informed consent (signed and dated) obtained before taking part in any trial-related activities.

Exclusion Criteria:

* Any current or previous disease, disorder, allergy or condition (including recent unexplained weight loss) that could affect the study conduct or laboratory assessments, or that presents undue risk from the study medication or procedures. Hypersensitivity to adhesive plasters or surgical tape.
* Any physical examination or screening investigation result that indicates the subject is unfit for the study.
* Scarring on upper arms, including extensive tattoos making skin reactions unevaluable.
* A positive virology test, urine test for drugs of abuse, or pregnancy test result (females of childbearing potential only).
* Recent use of prescribed or over-the-counter medication that, in the opinion of the Investigator or the Sponsor, will interfere with the study procedures or compromise safety.
* Received an investigational drug within 3 months (90 days) preceding patch application.
* Loss of ≥ 400 mL of blood (e.g. been a blood donor) within the past 3 months.
* Average weekly alcohol consumption of greater than 21 units (males) or 14 units (females), or habitually smokes ≥ 5 cigarettes or equivalent tobacco per day within the 6 months before patch application. Subjects may not smoke while confined to the study site. Subjects must not consume alcohol, or xanthine-containing foods or drinks within 48 hours prior to dosing until discharge.
* Lactating female subjects, and female subjects of childbearing potential who are not willing to use an acceptable form of contraception from the screening visit, during the study and for 90 days after the study.
* Employee of the Investigator or study centre, with direct involvement in the proposed study or other studies under the direction of that Investigator or study centre, as well as family members of the employees or the Investigator.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2010-03; Primary Completion 2010-04 (Actual); Study Completion 2010-04 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetic profile of the granisetron patch in healthy subjects when heat is applied | 0 - 196 hours post dose
  To assess the effect of locally applied heat on the pharmacokinetic profile of granisetron delivered from the patch. Subjects will be randomized to receive Treatment A Sancuso patch ONLY and Treatment B, Sancuso PLUS Cura-Heat pad. Sancuso will be worn by the subjects for 5 days continuously. The Cura-Heat pad will be applied over the patch for 4.5 hours on each of the 5 days. During these 5 days PK sampling is planned to measure the initial release of granisetron from the patch and cover the predicted maximum observed concentrations with or without the Cura-Heat pad in place.

SECONDARY OUTCOMES:
Safety and tolerability assessment | Up to 23 days post dose
  Safety and tolerability will be assessed by collection of adverse events, safety laboratory assessments, record of vital signs, conduct of physical examination and 12 lead ECG. In addition skin reaction at the patch and Cura-Heat pad application sites will be monitored.
residual granisetron after patch use in healthy subjects | 120 hours post dose
  • Residual granisetron after patch use and the calculation of in-vitro flux will be measured. All used patches will be returned to the manufacturer who will measure the amount of remaining granisetron in the patch and then the in-vitro flux will be calculated as follows: Amount delivered(assay amount-residual)/ number of days the patch was applied to the skin

CONTACTS AND LOCATIONS:
Overall Officials: Stuart J Mair, Principal Investigator — Quotient Clinical Limited
Locations (1):
- Quotient Clinical Limited, Edinburgh, United Kingdom